CLINICAL TRIAL: NCT05222022
Title: Engineering Evaluation of an Eye Movement Monitor Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. Light Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CLRT-001
Record Dates: First submitted 2022-01-11; First posted 2022-02-03 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: Eye movement measurement

STUDY DESIGN:
Intervention Model Description: Subjects participated in a design validation to evaluate the mechanism of action of the device to measure eye movement. This is not an applicable clinical trial to evaluate the effect of an intervention on biomedical or other health-related outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Design validation of mechanism of action of an eye movement measurement device (Experimental): Participants have retinal images captured with the Retitrack device to measure eye movements. The eye movement measurements are intended to validate the mechanism of action of the device.
  Interventions: Device: Retitrack

INTERVENTIONS:
Device: Retitrack — Retitrack device measures and analyzes eye movement

SUMMARY:
The objective of the engineering evaluation is to verify and validate the design of an eye movement monitor device, the Retitrack, for recording, viewing, measuring, and analyzing temporal characteristics of fixation and saccadic responses in human eyes when viewing a visual stimulus.

This engineering evaluation is not an applicable clinical trial. This is a design validation of the mechanism of action of the device to measure eye movement. This is not a clinical trial to evaluate the effect of an intervention on biomedical or other health-related outcomes.

DETAILED DESCRIPTION:
This non-significant risk device evaluation involves obtaining retinal images and eye movement measurements with the Retitrack device for purposes of design verification and validation testing. These measurements are not intended for use in diagnosing, preventing, monitoring, or alleviating a medical condition. This evaluation is not intended to assess biomedical or other health-related outcomes.

The evaluation involves the voluntary participation of up to 40 healthy adults who participate in a single device testing visit conducted over one or two days. The Retitrack is used to assess the alignment of the eye for image capture, the ability to measure and analyze eye movements for fixational and visually guided saccadic responses, and the usability of the device.

ELIGIBILITY:
Inclusion Criteria:

* History of good health
* Willing to participate in testing over 1 to 2 days with rest periods
* Willing to participate in device testing involving viewing visual targets, moving eyes as directed, and holding head steady
* Willing to have retinal images recorded for eye movement measurements

Exclusion Criteria:

* Refractive correction with glasses or contact lenses of more than 12 diopters of myopia or 4 diopters of hyperopia in either eye
* Active eye disease in either eye
* History of ocular surgery or ocular trauma in either eye within the past three months
* Ocular conditions in either eye that could interfere with obtaining a clear retinal image
* Ocular conditions in either eye that could affect the ability to view a stimulus or limit eye movement
* Neurological conditions that could affect eye movements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Device measurement of involuntary fixational microsaccade amplitude | 1 day (Single timepoint)
  Microsaccade amplitude (in degrees)
Device measurement of involuntary fixational microsaccade velocity | 1 day (Single timepoint)
  Microsaccade velocity (in degrees/second)
Device measurement of visually guided horizontal saccade amplitude | 1 day (Single timepoint)
  Horizontal saccade amplitude (in degrees)
Device measurement of visually guided horizontal saccade velocity | 1 day (Single timepoint)
  Horizontal saccade velocity (in degrees/second)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Theis, OD, Principal Investigator — Concussion Care Centre of Virginia, Ltd.
Locations (1):
- Blur Product Development, Cary, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No